CLINICAL TRIAL: NCT06006299
Title: Investigating the Feasibility of Using taVNS to Treat Insomnia in Individuals With Stage I-IV Breast Cancer
Brief Title: Investigating the Use of taVNS to Treat Insomnia in Individuals With Breast Cancer (taVNS-insomnia-BC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Alexandra Evancho, Assistant Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300010460; PREP grant (Other Grant/Funding Number: UAB Center for Palliative and Supportive Care)
Record Dates: First submitted 2023-07-31; First posted 2023-08-23 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer; Insomnia
Keywords: taVNS
MeSH Terms: conditions — Breast Neoplasms; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: All of the participants who are eligible will be in the taVNS group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- taVNS (Experimental): Participants will use the transauricular Vagus Nerve Stimulator provided to them by the lab for 14 days, 15 minutes prior to sleeping. Data will be collected via surveys, interviews, and Fitbit wear over the course of 2 months. A sleep diary will be kept to record sleep quality.
  Interventions: Device: transauricular Vagus Nerve Stimulation

INTERVENTIONS:
Device: transauricular Vagus Nerve Stimulation — Transcutaneous auricular vagus nerve stimulation (taVNS) is a form of transcutaneous electrical nerve stimulation (TENS) applied to peripheral nerves, considered a low-risk procedure. It involves the use of standard neurostimulation electrodes placed on the surface of the external ear. The taVNS method delivers low-intensity, pulsed electrical currents with a peak current amplitude of <4 mA, which is significantly lower than those used in most over-the-counter TENS devices for pain relief or muscle stimulation. By targeting the auricular branches of the vagus nerve, taVNS aims to stimulate specific neural pathways associated with various indications and intended uses. This non-invasive approach has broad applications in research, medical device treatments, health products, and cosmetic or lifestyle products.

SUMMARY:
In the present study, the investigators aim to investigate feasibility of utilizing noninvasive neuromodulation, specifically taVNS, as a nonpharmacologic approach to address insomnia in patients with stage I-IV breast cancer.

DETAILED DESCRIPTION:
The study will evaluate the feasibility, safety, and tolerability of nightly, at-home self-administered taVNS treatments. Study staff will monitor for adverse reactions, unanticipated adverse device events and severe adverse events as described to evaluate safety, tolerability, and biocompatibility. Additionally, investigators will estimate effect size by collecting outcome assessment data as described below. An additional objective is to use information gained through this study to inform product development activities. Specific information about the comfort, ease of use, and other user subject feedback will be used to inform future product development efforts for optimizing device designs.

Specific Aim 1: To evaluate the feasibility of using taVNS for patients with breast cancer to treat insomnia. HYPOTHESIS: Investigators expect that 40 patients with stage I-III breast cancer and insomnia will be enrolled and undergo taVNS to address insomnia, quantified by various sleep related outcome measures, with an estimated recruitment rate of 70%, eligibility rate of 70%, completion rate of 80%, and follow up rate of 80%.

Specific Aim 2: To evaluate the efficacy of repeated, nightly taVNS on sleep quality, anxiety, and cancer related fatigue. HYPOTHESIS: Investigators hypothesize that patients will report improved sleep, anxiety, depression, and cancer related fatigue after one week of taVNS.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years of age
2. diagnosed stage I-IV breast cancer
3. self-reported difficulty falling asleep, staying asleep, or waking up too early, for at least three nights per week for a duration of at least three months
4. beginning or worsening of sleep disturbance since cancer diagnosis (did your sleep problems begin or get worse with the diagnosis of cancer or with chemotherapy?)
5. English-speaking

Exclusion Criteria:

1. Are using a daily sleep aid except melatonin (use of a sleep aid as needed will be permitted, and use will be noted).
2. have a history of severe mental illness
3. have an implanted medical device of any type
4. have a history of seizures
5. have peripheral neuropathy including temporal mandibular disorders and Bells Palsy
6. have vasovagal syncope
7. have moderate to severe cognitive impairment
8. have <6 months to live as determined by the physician

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-09-26 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Feasibility of using transauricular Vagus Nerve Stimulation to treat insomnia in individuals with stage I-IV breast cancer. | 2 months
  Our mixed method approach for evaluating feasibility includes measuring eligibility rates, retention rates, refusal rates, and follow-up rates as well as analyzing information gathered from interviews. In this feasibility study, a recruitment rate of at least 70% within 6 weeks, an eligibility rate of >70%, a completion rate of 80% of the protocol, and a follow up rate of 80% will be considered successful.

SECONDARY OUTCOMES:
Insomnia Severity Index | 2 months
  The Insomnia Severity Index (ISI) is a seven-question survey that is commonly used to identify and quantify the severity of insomnia over the past 2 weeks. Using a five-point Likert-type scale, it asks questions regarding difficulty falling asleep and maintaining sleep, satisfaction with sleep, noticeability of sleep disturbances, and distress. Out of total possible score of 28, a score of 8 is generally regarded as the optimal cut-off for clinical significance and a score of 15 indicates chronic insomnia syndrome.
The Pittsburgh Sleep Quality Index (PSQI) | 2 months
  The Pittsburgh Sleep Quality Index (PSQI) is a widely used self-report questionnaire designed to assess sleep quality and disturbances in individuals. It is a valuable tool in evaluating the severity of insomnia and other sleep-related issues.
  The PSQI generates a total score that ranges from 0 to 21, with higher scores indicating poorer sleep quality. A lower PSQI score suggests better sleep quality and fewer sleep disturbances, while a higher score implies more significant sleep problems and reduced overall sleep satisfaction. The index considers various aspects of sleep, including sleep latency, sleep duration, sleep efficiency, sleep disturbances, use of sleep medications, and daytime dysfunction. The score helps to quantify and categorize individuals' sleep patterns, enabling healthcare professionals to identify sleep-related issues and develop appropriate interventions to improve sleep quality and overall well-being.
Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Assessment (Short Form) | 2 months
  The PROMIS Anxiety Assessment Short Form is a concise and validated self-report questionnaire used to evaluate anxiety symptoms in individuals. It is part of the Patient-Reported Outcomes Measurement Information System (PROMIS) toolset, widely recognized for assessing various health-related aspects.
  The PROMIS Anxiety Assessment Short Form generates a score that reflects the severity of anxiety symptoms experienced by an individual. The score is standardized, with higher values indicating higher levels of anxiety. Conversely, lower scores represent less severe anxiety symptoms. By utilizing this assessment, healthcare professionals can quantify and monitor anxiety levels in patients, aiding in the identification of anxiety-related issues and facilitating personalized interventions for improved mental well-being.
Generalized Anxiety Disorder 7 (GAD-7) | 2 months
  The GAD-7 generates a total score ranging from 0 to 21, with higher scores indicating higher levels of anxiety symptom severity. The score is typically interpreted as follows:
  0 to 4: Minimal anxiety 5 to 9: Mild anxiety 10 to 14: Moderate anxiety 15 to 21: Severe anxiety
  A lower GAD-7 score suggests minimal to mild anxiety, while higher scores indicate moderate to severe anxiety symptoms. Healthcare professionals utilize the GAD-7 to assess and monitor anxiety levels in individuals, helping to guide treatment decisions and interventions aimed at improving mental well-being and overall quality of life.
Patient Health Questionnaire-9 (PHQ-9) | 2 months
  The PHQ-9 generates a total score ranging from 0 to 27, with higher scores indicating higher levels of depressive symptom severity. The score is typically interpreted as follows:
  0 to 4: Minimal or no depression 5 to 9: Mild depression 10 to 14: Moderate depression 15 to 19: Moderately severe depression 20 to 27: Severe depression
  A lower PHQ-9 score suggests minimal or no depression, while higher scores indicate varying degrees of depressive symptoms. Healthcare professionals use the PHQ-9 to assess and monitor depression levels in individuals, facilitating treatment decisions and interventions aimed at improving mental well-being and overall quality of life.
Cancer Fatigue Scale (CFS) | 2 months
  The Cancer Fatigue Scale (CFS) is a self-report questionnaire designed to assess an individual's sense of fatigue in the context of cancer-related fatigue. The questionnaire consists of 15 questions, and participants are asked to rate their current state of fatigue on a scale from 1 (No) to 5 (Very Much). The scale measures three different aspects of fatigue: physical, affective, and cognitive.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Evancho, DPT, Principal Investigator — The University of Alabama at Birmingham
Locations (2):
- United States (2):
  - UAB Lakeshore Collaborative (WHARF), Birmingham, Alabama
  - UAB Spain Rehabilitation Center, Birmingham, Alabama

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Do M, Evancho A, Tyler WJ. Bilateral transcutaneous auricular vagus nerve stimulation for the treatment of insomnia in breast cancer. Sci Rep. 2025 Dec 4;16(1):1081. doi: 10.1038/s41598-025-30600-6. PMID 41345210